CLINICAL TRIAL: NCT01701726
Title: Acupuncture for Patients With Mild Hypertension: Study Protocol of an Open-label Multicenter Randomized Controlled Trial
Brief Title: Effect of Acupuncture on Patients With Mild Hypertension
Acronym: EAPMH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012CB518501-1
Record Dates: First submitted 2012-09-26; First posted 2012-10-05 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension; Acupuncture; Specificity; Acupoints effect; randomized controlled trials
MeSH Terms: conditions — Essential Hypertension | interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupuncture (Experimental): Two types of acupuncture are given, one is acupuncture at affected meridian points, the other is at non-affected. For the first type, We select the acupoints from the affected meridians.Patients in this group are divided into two subgroups according meridian syndrome differentiation(jue-yin style,yang-ming style).Patients pertaining to Jue-yin-style are treated with taichong (LR3), renying(ST9), taixi(KI3), neiguan(PC6) .Patients pertaining to Yang-ming-style: taichong(LR3), renying(ST9), zusanli(ST36), quchi(LI11). For the second,We select the acupoints from the non-affected meridians.Patients assigned into the non-affected meridian acupuncture group will be treated with Fengchi (GB20), waiguan(SJ5), yinlingquan(SP9), xuehai (SP10).
  Interventions: Other: acupuncture
- Sham acupuncture (Sham Comparator): we use sham acupoints:
  1. The edge of the tibia (1-2cm lateral and horizontal to the zusanli (ST36))
  2. Half way between the tip of the elbow and the axilla
  3. On the ulnar side of the arm, half way between the epicondylus medialis of the humerus and the ulnar side of the wrist.
  4. 2cm superior to fu tu(LI18)
  Interventions: Other: Sham acupuncture
- Waiting list (No Intervention): Participants who will be randomized into the waiting-list group will not receive any acupuncture treatment throughout 13-week observation period. At the end of trial, if the participant would like to be treated with acupuncture, it will be provided three times weekly for 6 weeks.

INTERVENTIONS:
Other: acupuncture — In each session, acupuncture are applied bilaterally. Except the acupoints around the neck(ST9.GB20.non-acupoints 4) ,6 auxiliary needles will be punctured at 2mm lateral to each acupoints or non-acupoints.as to auxiliary needle we will not do any manipulation. We use transcutaneous electric acupoints stimulation to stimulate the acupoints and non-acupoints.
  Other Names: electroacupuncture
  Arms: Acupuncture
Other: Sham acupuncture — In contrast to acupuncture, sham acupuncture is given at 4 sham points with skin penetration. Electroacupuncture is also applied.
  Arms: Sham acupuncture

SUMMARY:
This is a large scale, open-label, multicenter, randomized controlled clinical trial with four parallel arms. This trial aims to evaluate the effectiveness of affected meridian acupuncture for patients with mild hypertension,with respect to decreasing their blood pressure, safety of acupuncture ,and improving their quality of life as well.

DETAILED DESCRIPTION:
Investigators plan to recruit 428 hypertensive patients. Eligible patients will be randomized to four different groups.ⅰ. the affected meridian acupuncture group (AMA, n=107) will be treated with acupoints on affected meridians.ⅱ.the non-affected meridian acupuncture group (NMA, n=107) will be treated with acupoints on non-affected meridians.ⅲ.invasive sham acupuncture group(ISA, n=107)will be provided with sham acupoints treatment.ⅳ.waiting-list group(WL, n=107)will not be given any intervention.

ELIGIBILITY:
Inclusion Criteria：

1. Patients whose age between 40 and 75 years old, male and female;
2. Patients who meet the diagnostic criteria of mild hypertension according to JNC-7 and China's prevention and cure guide of hypertension. mild hypertension (WHO/ISH criteria stage I) Systolic blood pressure 159≥(SBP) ≥140 and/or diastolic blood pressure 99≥(DBP) ≥90 .
3. Patients who are initially diagnosed as mild hypertension or have been diagnosed as mild hypertension before but have not taken any antihypertensive drugs.
4. Patients who are diagnosed as yue-yin style (yin-deficiency accompany with hyperactivity of yang) or yang-ming style (obstruction of phlegm and dampness) according to meridian syndrome differentiation
5. Patients who have a good understanding of our study. and willing to comply with our study protocol.
6. Informed consent form must be signed by patient or lineal relative.
7. All the tips are matched will be included.

Exclusion Criteria:

1. Patients who have been diagnosed as secondary hypertension or malignant hypertension(e.g. Cushing's syndrome, coarctation of the aorta，phaeochromocytoma, renal parenchymal disease，primary aldosteronism， renovascular hypertension, obstructive sleep apnoea，drug induced hypertension et al )
2. Patients who accompany with other severe medical conditions (e.g. endocrine disorders, cardiovascular disease. Digestive disease. hepatic dysfunction，cerebral vascular disease. renal disease. haematologic disease et al). Who may be not safe to join our study.
3. Patients with a chronic disease which might not suitable for our study. e.g: epilepsy ,severe depression or anxiety (SAS≥70,SDS≥70) ,psychosis, allergic constitution, accompany with any infection.
4. Pregnant women or women in lactation or women of child bearing potential plan to conceive in the recent six months.
5. Patients who currently participate in another clinical trial.
6. Patients who Had been treated with acupuncture during the previous three months
7. If one of the tips mentioned above is matched will be excluded.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2012-07; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Average systolic and average diastolic blood pressure by 24-hour ambulatory blood pressure monitoring | 6weeks after randomization.
  The primary outcome is the average systolic and average diastolic blood pressure measured at 6 weeks after randomization by 24-hour ambulatory blood pressure monitoring.
Visit-to-visit blood pressure variation | 6 weeks after randomization
  Assessed by 24-hour ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Average systolic and average diastolic blood pressure during the daytime and nighttime. | 0 day, 6weeks, 9weeks, 12weeks after randomization.
  The daytime is from 8AM to 10PM,nighttime is 10PM -8AM.
Average systolic and average diastolic blood pressure during the daytime and nighttime. | 0 day, 6weeks, 9weeks, 12weeks after randomization.
  The daytime is defined as 8AM-10PM.Nighttime is defined as 10PM -8AM.
changes in patients health-related quality of life | 0 day and 6 weeks after randomization.
  SF-36 (Medical Outcomes Study 36-Item Short Form)questionnaire Chinese version. The scale contains eight dimensions (physical function, role physical, bodily pain, general health, vitality, social function, role emotional, mental health) and two summary components (physical and mental ),scale 0-100.lower scores indicate poorer quality of life.
Adverse events | 0 day, 6weeks, 9weeks, 12weeks after randomization
  Adverse events are defined as any unexpected or discomfort signs, symptoms or diseases, regardless of the intervention. If any adverse events happen during the entire observation period, all the details should be documented in the case report form. These adverse events include bleeding, hematoma, fainting, serious pain, and local infection.

CONTACTS AND LOCATIONS:
Overall Officials: fan-rong Liang, MD, Study Chair — Chengdu University of Tranditional Chinese Medicine
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Wang JM, Yang MX, Wu QF, Chen J, Deng SF, Chen L, Wei DN, Liang FR. Improvement of intestinal flora: accompany with the antihypertensive effect of electroacupuncture on stage 1 hypertension. Chin Med. 2021 Jan 7;16(1):7. doi: 10.1186/s13020-020-00417-8. PMID 33413552
- [Derived] Li J, Zheng H, Zhao L, Li Y, Zhang Y, Chang XR, Wang RH, Shi J, Cui J, Huang YL, Li X, Chen J, Li DH, Liang FR. Acupuncture for patients with mild hypertension: study protocol of an open-label multicenter randomized controlled trial. Trials. 2013 Nov 11;14:380. doi: 10.1186/1745-6215-14-380. PMID 24216113